CLINICAL TRIAL: NCT05337735
Title: A Phase II Clinical Trial to Evaluate Safety and Efficacy of XmAb20717 in Advanced Rare Cancers
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0589; NCI-2022-02841 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-28; First posted 2022-04-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Microsatellite High Cancers; Peritoneal Mesothelioma; Extrapulmonary High Grade; Neuroendocrine Carcinomas; Cervical Carcinoma; Hodgkin's Lymphoma; Pleural Mesothelioma; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Uterine Cervical Neoplasms; Hodgkin Disease; Mesothelioma, Malignant; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- XmAb20717 (Experimental): Participants will receive XmAb20717 by vein over 1 hour on Days 1 and 15 of each cycle.
  Interventions: Drug: XmAb20717

INTERVENTIONS:
Drug: XmAb20717 — Given by vein (IV)

SUMMARY:
To test the safety of and effectiveness of XmAb20717 for participants with advanced rare cancers.

DETAILED DESCRIPTION:
Primary Objective:

Efficacy of XmAb20717 as defined by objective response (defined as a complete response [CR] or partial response [PR] on two consecutive occasions ≥4 weeks apart) as determined by an independent radiologist according to RECIST v1.1 (modified RECIST for pleural mesothelioma)

Secondary Objectives:

1. Objective response as determined by an independent radiologist according to immune-modified RECIST
2. Progression-free survival (PFS) (defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first) as determined by an independent radiologist according to RECIST v1.1 (modified RECIST for pleural mesothelioma).
3. Duration of response (DoR) (defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first) as determined by an independent radiologist according to RECIST v1.1 (modified RECIST for pleural mesothelioma)
4. Disease control as determined by an independent radiologist according to RECIST v1.1 (modified RECIST for pleural mesothelioma)
5. Overall survival (OS) (defined as the time from enrollment to death from any cause)
6. PFS as determined by an independent radiologist according to immune-modified RECIST
7. DoR as determined by an independent radiologist according to immune-modified RECIST
8. Disease control as determined by an independent radiologist according to immune-modified RECIST
9. Occurrence and severity of AEs, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

Exploratory Objective

To identify biomarkers that are predictive of response and/or are associated with progression to a more severe disease state (i.e., prognostic biomarkers).

ELIGIBILITY:
Study Participant Inclusion Criteria

Inclusion Criteria:

1. Is able to complete signed informed consent. Patients for whom English is not their primary language are eligible for participation with translator assistance during the informed consent process.
2. Is of age ≥ 18
3. Is able, in the investigator's judgment, to comply with the study protocol
4. Has measurable disease according to RECIST v1.1 The pleural mesothelioma cohort will require measurable disease according to either modified RECIST or RECIST; the Hodgkin lymphoma patients will be assessed by the 2014 Lugano criteria (see Appendix F)
5. Has an ECOG performance status of 0 - 1
6. Has adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

   * ANC ≥ 1.0×109/L without granulocyte colony-stimulating factor support (for the lymphoma cohort only, Absolute neutrophil count of ≥ 1.0×109/L without growth factor support for 3 days prior to screening assessment.)
   * Lymphocyte count ≥ 0.5×109/L
   * Platelet count ≥ 100× 109/L without transfusion (for the lymphoma cohort only: platelet count of ≥ 50×109/L without transfusion for 3 days prior to screening assessment)
   * Hemoglobin ≥ 90 g/L (for the lymphoma cohort only: Hemoglobin >80 g/L without transfusion for 3 days prior to screening assessment) (For platelet count and hemoglobin, patients may be transfused to meet either criterion but not within 14 days prior to initiation of study treatment)
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5× upper limit of normal (ULN), with the following exceptions:
   * Patients with documented liver metastases: AST and ALT ≤ 5×ULN
   * Patients with documented liver or bone metastases: ALP ≤ 5×ULN
   * Serum bilirubin ≤ 1.5 ×ULN with the following exception:
   * Serum creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) ≥50 mL/min OR 24-hour urine creatinine clearance ≥50 mL/min
   * Serum albumin ≥ 2.5 g/dL
   * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5×ULN
   * For patients receiving therapeutic anticoagulation: is on a stable anticoagulant regimen without changes in agent and / or dose in the past 30 days
7. Must agree to use a highly effective method of birth control (as defined in Section 7.4.1) (female patients and male patients with female partners of childbearing potential) during and for 6 months after last dose of study treatment. Also see related information in Section 6.6.10.8.

   .

Basket-specific Inclusion Criteria:

1. Peritoneal Mesothelioma: Has advanced MPeM that was previously treated with and refractory/intolerant to platinum-pemetrexed systemic chemotherapy or has not received treatment and is ineligible for platinum-pemetrexed treatment
2. Pleural Mesothelioma: Has unresectable MPM and is treatment naïve or has received any line of prior therapy, including anti-PD1/anti-PDL1/anti-CTLA4.
3. High-grade Neuroendocrine Carcinoma: Has extra-pulmonary site carcinoma (small-cell- and large-cell lung cancer excluded) and has received therapy with a platinum-based chemotherapy regimen
4. MSI-H Cancers: Has not had anti-PD1 / anti-PDL1 / anti-CLTA4 therapyMSI-H/dMMR, locally advanced or metastatic solid tumors. Locally advanced solid tumors are defined by having ≥20% chance of recurrence with surgery alone. Patients with localized solid tumors are also eligible if they have a high risk for surgical mortality defined as >5% by ACS National Surgery Quality Improvement Program. Patients being treated with neoadjuvant intent may be treated for up to 6 months prior to surgical resection, though in patients with clear clinical benefit as deemed by treating physicians, a non-operative approach-treatment duration ≥ 6 months (and up to 2 years)-may be considered.

   Note: ASC = American College of Surgeons, MSI-H = microsatellite instability-high, dMMR = deficient mismatch repair.
5. Lymphoma: Has relapsed, refractory classical Hodgkin lymphoma and has received first-line chemotherapy. Prior treatment with anti-PD1 / PDL1 antibody is not exclusionary.
6. Cervical Cancer: Has recurrent, metastatic, or persistent cervical cancer (squamous cell carcinoma, adenosquamous, or adenocarcinoma of the cervix) and has received at least one prior line of systemic therapy and not amenable to curative treatment. Prior treatment with anti-PD1 / PDL1 antibody is not exclusionary.
7. Small-cell lung cancer: Extensive-stage small-cell lung cancer following treatment with prior platinum-based therapy, which can include prior anti-PD1, anti-PDL1, but not anti-CTLA4.

Study Participant Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

1. Received treatment for the studied cancer within 21 days prior to initiation of study treatment
2. Received treatment with targeted therapies or investigational therapies within 21 days or for the duration of 5 half-lives prior to initiation of study treatment
3. Has a history of severe allergic, anaphylactic, or other hypersensitivity reactions to study drug
4. Has active known- or suspected autoimmune disease (allowed are patients with vitiligo; type 1 diabetes mellitus, or residual hypothyroidism due to an autoimmune condition that is treatable with hormone-replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and non-steroidal anti-inflammatory drugs).
5. Has any condition that requires systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of study drug (except that inhaled or topical corticosteroids or brief courses of corticosteroids given for prophylaxis of contrast dye allergic response are permitted).
6. Has a history or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary-, renal-, metabolic-, hematologic-, or psychiatric-) other than their primary malignancy, that in the opinion of the Investigator would pose a risk to patient safety or interfere with study evaluations, procedures, or completion.
7. Has had any serious bacterial, viral, parasitic, or systemic fungal infections within 14 days prior to the first dose of study drug.
8. Received prior treatment with any checkpoint-inhibitor therapy regimen that targets PD1/PDL1 or CTLA-4 (this does not apply to candidates for the lymphoma, pleural mesothelioma, cervical cancer or SCLC cohorts-see basket-specific inclusion criteria).
9. Received a live-virus vaccine within 30 days prior to first dose of study drug (vaccines that do not contain live virus are permitted).
10. Has another malignancy, except for non-melanoma skin cancer, in situ cervical cancer, or bladder cancer (Tis and T1) that has been adequately treated during the 3 years prior to screening (Note: For MSI-H cohort, prior history of malignancies are allowed unless this may be a competing risk for mortality while on study per the investigator).
11. Has untreated or unstable brain metastases. Allowed are those with known brain metastases who have been previously treated and are asymptomatic. If prior local therapy was received, it must have been completed at least 14 days prior to receiving study drug.
12. Has evidence of current ILD or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids
13. Is breastfeeding or plans to initiate breastfeeding during the study treatment or within 6 months of taking study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To establish the efficacy of XmAb20717 as measured by overall response rate. | through study completion, an average of 1 year
  Number of Participants With Objective Radiographic response as Assessed by RECIST v.1.1

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Nageshwara Dasaru, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org